CLINICAL TRIAL: NCT04799210
Title: Human Factors Actual-Use Confirmatory Validation Study of the Eximis CS (Contained Segmentation) System ("Contain" Study)
Brief Title: Human Factors Actual-Use Clinical Protocol
Acronym: CONTAIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device performance was not as anticipated.
Sponsor: Eximis Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP2020-001
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Laparoscopic Gynecological Surgery
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Human Factors Actual Use (Experimental): Confirm device use safety and effectiveness of the Eximis CS (Contained Segmentation) System in actual use
  Interventions: Device: Eximis CS (Contained Segmentation) System

INTERVENTIONS:
Device: Eximis CS (Contained Segmentation) System — Containment, segmentation and extraction of uterine tissue in pre-menopausal women undergoing laparoscopic hysterectomy or myomectomy for non-cancer indications.
  Other Names: Eximis CS; EX-900K-CLIN

SUMMARY:
The purpose of this study is to confirm device use safety and effectiveness of the Eximis CS (Contained Segmentation) System in actual use by representative users, use, and use environments as required for regulatory agency clearance for commercial use.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm study to confirm device use safety and effectiveness in an actual use setting when utilized by gynecological surgeons during surgery for containment, segmentation and extraction of uterine tissue in pre-menopausal women undergoing laparoscopic hysterectomy or myomectomy for non-cancer indications.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 21 and < 50 years.
2. Planned laparoscopic hysterectomy or myomectomy.
3. Tissue specimen is <11 cm in maximum diameter based on standard preoperative assessment.
4. Pre-operative evaluation which may include imaging, cervical cancer screening, and endometrial biopsy has been completed.
5. Signed informed consent.
6. Willing to adhere to protocol requirements and complete follow-up.

Exclusion Criteria:

1. Subject is post-menopausal, defined as amenorrhea >12 months in the absence of ovulation suppression.
2. Known or suspected malignancy of gynecological origin as determined by standard clinical practice.
3. Candidate for en bloc tissue removal, for example through the vagina or via a mini-laparotomy incision.
4. Hemoglobin < 8 g/dl within 30 days prior to surgery.
5. Subject has a current history of undiagnosed genital bleeding.
6. Subject has an implanted electronic device where use of radiofrequency (RF) energy would be contraindicated (e.g., pacemaker, internal defibrillator).
7. Medical condition, surgical history, or intra-operative findings, which in the option of the investigator, precludes utilization of the Eximis CS System.
8. Known allergy to polyurethane, polyethylene, thermoplastic fluoropolymer and/or chlorinated polyvinyl chloride.
9. Concurrent participation in another therapeutic or interventional clinical trial with investigational pharmaceutical agent(s) or medical device(s) that could impact evaluation of this study as determined by the Investigator.
10. Inability to comply with the study procedures or follow-up in the opinion of the investigator.
11. Subject is pregnant.
12. Intraoperative Exclusion: Abdominal wall thickness at the umbilicus incision site is > 8 cm.

Ages: 21 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pre-menopausal women undergoing laparoscopic hysterectomy or myomectomy for non-cancer indications.
Enrollment: 3 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
The number of procedures where all critical tasks related to the Eximis CS are performed without serious use error. | Through study completion, anticipated to be 4-6 months
  Primary Endpoint

SECONDARY OUTCOMES:
Number of procedures successfully completed with use of the Eximis CS device. | Through study completion, anticipated to be 4-6 months
  Secondary Endpoint
Number of Capture Bags with breach of containment. | Through study completion, anticipated to be 4-6 months
  Secondary Endpoint
The number and severity of user adverse events caused by use error. | Day of surgery
  Secondary Endpoint
The number and severity of subject adverse events caused by use error. | Minimum 30 days (Standard of care follow-up 4-6 weeks)
  Secondary Endpoint
All other adverse events. | Minimum 30 days (Standard of care follow-up 4-6 weeks)
  Secondary Endpoint

OTHER OUTCOMES:
Duration of the segmentation/extraction procedure (from insertion of the Eximis CS deployment instrument into the abdomen until removal of the Eximis CS Capture Bag from the abdomen). | Day of surgery
  For Informal Evaluation
Duration of the surgical procedure (from skin incision to skin closure). | Day of surgery
  For Informal Evaluation
Length of incision (mm) used for the Eximis CS device at procedure end (removal of Eximis CS Capture Bag). | Day of surgery
  For Informal Evaluation
Removed tissue weight (grams). | Day of surgery
  For Informal Evaluation
Number of extracted tissue segments per subject. | Day of surgery
  For Informal Evaluation
The size (mm) of the largest segment will be recorded, defined as the segment with the largest cross-sectional area of the surface that is parallel with the incision opening. | Day of surgery
  For Informal Evaluation
Subject's pathology results of the extracted tissue and pathologist assessment of radiofrequency (RF) energy impact to the tissue, if any, from use of the Eximis CS device. | Day of surgery
  For Informal Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Sawsan As-Sanie, MD, MPH, Principal Investigator — Women's Hospital, University of Michigan
Locations (7):
- United States (7):
  - Advanced Women's Health Institute, Greenwood Village, Colorado
  - AdventHealth Medical Group Gynecologic Surgery at Celebration, Celebration, Florida
  - Swor Women's Care, Sarasota, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - Advanced Gynecologic Surgery Institute, Park Ridge, Illinois
  - University of Michigan Health System, Ann Arbor, Michigan
  - ProMedica Health System, Sylvania, Ohio

IPD SHARING:
Plan to Share IPD: No